CLINICAL TRIAL: NCT02258347
Title: Use of a High Intensity Focused Ultrasound (HIFU) in Patients With Non-malignant Thyroid Nodules.
Brief Title: HIFU in Patients With Non-malignant Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/REG/NT
Record Dates: First submitted 2014-09-26; First posted 2014-10-07 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2018-05

CONDITIONS: Non-malignant Thyroid Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse

SUMMARY:
Use of a high intensity focused ultrasound (HIFU) in patients with non-malignant thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years or older.
* Patient presenting with at least one thyroid nodule with no signs of malignancy:

  1. Non suspect clinically and at ultrasonography imaging
  2. Benign cytological diagnosis at fine-needle aspiration biopsy (FNAB) from the last 6 months
  3. Normal serum calcitonin
  4. No history of neck irradiation
* Normal thyroid-stimulating hormone (TSH).
* Targeted nodule accessible and eligible to HIFU
* Absence of abnormal vocal cord mobility at laryngoscopy.
* Nodule diameter ≥ 10mm measured by ultrasound.
* Nodule volume inferior to 10 cc
* Composition of the targeted nodule(s) : no more than 30% cystic

Exclusion Criteria:

* Head and/or neck disease that prevents hyperextension of neck.
* Known history of thyroid cancer or other neoplasias in the neck region.
* History of neck irradiation.
* Macrocalcification inducing a shadow in the thyroid significant enough to preclude the HIFU treatment
* Posterior position of the nodule if the thickness of the nodule is <15mm
* Pregnant or lactating woman
* Any contraindication to the assigned analgesia/anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2015-10-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of thyroid nodule's volume changes following HIFU therapy assessed by ultrasonography (US) | Month 6 and Month 12
Evaluation of thyroid nodule's structure changes following HIFU therapy assessed by ultrasonography (US) | Month 6 and Month 12
Evaluation of thyroid nodule's vascularisation changes following HIFU therapy assessed by ultrasonography (US) | Month 6 and Month 12

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Day 1, Month 1, Month 3, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Frasoldati, Dr, Principal Investigator
Locations (1):
- Istituto in tecnologie avanzate e modelli assistenziali in oncologia, Reggio Emilia, Italy